CLINICAL TRIAL: NCT04460391
Title: Influence of Early Standing Training on ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Ph.D., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intensive rehabilitation
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Early standing training and routine rehabilitation
  Interventions: Behavioral: Intensive rehabilitation
- control group (Active Comparator): Conventional rehabilitation，Muscle training and breathing training
  Interventions: Behavioral: Intensive rehabilitation

INTERVENTIONS:
Behavioral: Intensive rehabilitation — Early standing training and routine rehabilitation

SUMMARY:
Influence of early standing training on ICU patients

DETAILED DESCRIPTION:
Objective: To study the effect of early standing training on ICU patients.Background: Early severe rehabilitation is of great significance for patients, which can help patients withdraw from mechanical ventilation as soon as possible, improve pulmonary ventilation, and promote early walking.However, patients on mechanical ventilation are more prone to delirium, muscle weakness, ventilator dependence and other problems. Early standing training can significantly improve patients' lower limb muscle strength, improve diaphragm function, improve the prognosis of patients, and reduce the length of hospital stay.Methods: selecting stable hemodynamics in ICU patients with mechanical ventilation, randomly divided into two groups, a group of routine rehabilitation training, another group stand for regular rehabilitation and early training, with the aid of electric beds, on the first day of patients, to evaluate the seventh day, the 14th day, and collect the basic information for patients and strength assessment, blood gas analysis, the diaphragm of the bed and ultrasound and muscle ultrasound, and record the patient's mortality within 28 days, the incidence of delirium, decannulation rate, etc., recorded in patients with mechanical ventilation time and the time required to walk independently and ICU stay time.

ELIGIBILITY:
Inclusion Criteria:

* The age is ≥ 18 years old;
* the hemodynamics is stable;
* 50 < heart rate < 120 beats / min ;
* 90 < systolic blood pressure < 200mmHg ;
* 55 < mean arterial pressure < 120mmHg;
* do not increase the dose of pressor drugs for at least 2 hours;
* intracranial pressure is stable and there are no seizures within 24 hours;
* the respiratory state is stable;
* the patient's finger pulse oxygen saturation ≥ 88%;
* Oxygen concentration less than 60%；
* Terminal positive expiratory pressure<12cmH2O；
* 10 < respiratory frequency < 35 beats / min.

Exclusion Criteria:

* Pregnancy;
* acute cardio-cerebrovascular events;
* spinal or limb fractures;
* active bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Medical Research Council | day 1
  Muscle strength assessment of ICU patients，Out of 60 points，Less than 48 points had acquired muscle weakness in the ICU.
Medical Research Council | day 7
  Muscle strength assessment of ICU patients，Out of 60 points，Less than 48 points had acquired muscle weakness in the ICU.
Medical Research Council | day 14
  Muscle strength assessment of ICU patients，Out of 60 points，Less than 48 points had acquired muscle weakness in the ICU.
Berg Balance Scale | day 1
  Balance grade score,The highest 56 points,The higher the score, the better the balance.
Berg Balance Scale | day 7
  Balance grade score,The highest 56 points,The higher the score, the better the balance.
Berg Balance Scale | day 14
  Balance grade score,The highest 56 points,The higher the score, the better the balance.
FIM Function Independent Scale | day 1
  Functional independence assessment,The lowest score is 18 and the highest is 126,The higher the score, the more independent it is.
FIM Function Independent Scale | day 7
  Functional independence assessment,The lowest score is 18 and the highest is 126,The higher the score, the more independent it is.
FIM Function Independent Scale | day 14
  Functional independence assessment,The lowest score is 18 and the highest is 126,The higher the score, the more independent it is.
Holden walk classification | day 1
  Levels 0 to 5,The higher the grade, the better the ability to walk
Holden walk classification | day 7
  Levels 0 to 5,The higher the grade, the better the ability to walk
Holden walk classification | day 14
  Levels 0 to 5,The higher the grade, the better the ability to walk
arterial blood gas analysis | day 1
  PH,normal range 7.35-7.45
arterial blood gas analysis | day 7
  PH,normal range 7.35-7.45
arterial blood gas analysis | day 14
  PH,normal range 7.35-7.45
partial pressure of carbon dioxide | day 1
  normal range 35-45 mmHg
partial pressure of carbon dioxide | day 7
  normal range 35-45 mmHg
partial pressure of carbon dioxide | day 14
  normal range 35-45 mmHg
oxygenation index | day 1
  Normal adults are 400,the higher，the better
oxygenation index | day 7
  Normal adults are 400,the higher，the better
oxygenation index | day 14
  Normal adults are 400,the higher，the better
lactic acid | day 1
  normal range 0.5-1.6mmol/L
lactic acid | day 7
  normal range 0.5-1.6mmol/L
lactic acid | day 14
  normal range 0.5-1.6mmol/L
Diaphragmatic movement | day 1
  The distance the diaphragm moves downward during inhalation,Normal adults are 1.4cm.
Diaphragmatic movement | day 7
  The distance the diaphragm moves downward during inhalation,Normal adults are 1.4cm.
Diaphragmatic movement | day 14
  The distance the diaphragm moves downward during inhalation,Normal adults are 1.4cm.
Diaphragm contraction rate | day 1
  Normal adults are 1.3cm/s
Diaphragm contraction rate | day 7
  Normal adults are 1.3cm/s
Diaphragm contraction rate | day 14
  Normal adults are 1.3cm/s
Diaphragm thickness at end of breath | day 1
  Normal adults are 0.15cm
Diaphragm thickness at end of breath | day 7
  Normal adults are 0.15cm
Diaphragm thickness at end of breath | day 14
  Normal adults are 0.15cm
Diaphragm thickness at end of inhalation | day 1
  Normal adults are 0.28cm
Diaphragm thickness at end of inhalation | day 7
  Normal adults are 0.28cm
Diaphragm thickness at end of inhalation | day 14
  Normal adults are 0.28cm
Diaphragmatic thickness variation rate | day 1
  Less than 20% have diaphragmatic dysfunction
Diaphragmatic thickness variation rate | day 7
  Less than 20% have diaphragmatic dysfunction
Diaphragmatic thickness variation rate | day 14
  Less than 20% have diaphragmatic dysfunction
E-T index | day 1
  Product of inspiratory time and diaphragmatic mobility,The higher the extubation success rate, the higher the extubation success rate.
E-T index | day 7
  Product of inspiratory time and diaphragmatic mobility,The higher the extubation success rate, the higher the extubation success rate.
E-T index | day 14
  Product of inspiratory time and diaphragmatic mobility,The higher the extubation success rate, the higher the extubation success rate.
Timed Inspiration | day 1
  Normal adults are 1s
Timed Inspiration | day 7
  Normal adults are 1s
Timed Inspiration | day 14
  Normal adults are 1s
Rectus femoris thickness | day 1
  The thicker the muscle, the better
Rectus femoris thickness | day 7
  The thicker the muscle, the better
Rectus femoris thickness | day 14
  The thicker the muscle, the better
Thickness of tibialis anterior muscle | day 1
  The thicker the muscle, the better
Thickness of tibialis anterior muscle | day 7
  The thicker the muscle, the better
Thickness of tibialis anterior muscle | day 14
  The thicker the muscle, the better

SECONDARY OUTCOMES:
Mechanical ventilation time | three months
  Mechanical ventilation time
icu length of stay | three months
  icu length of stay
Time required for independent walking | three months
  Time required for independent walking
delirium | 28 days
  Confusion Assessment Method of the Intensive Care Unit. Positive is delirium.
mortality | 28 days
  mortality
reintubation | 28 days
  Note whether intubation was performed within 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: xin li xie, Principal Investigator — The First Medical Center of PLA General Hospital